CLINICAL TRIAL: NCT00233649
Title: DIALOOG: Crestor in Patients With Diabetes Mellitus Type 2: Lowering of LDL-C Levels to New European Guidelines
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NL401017
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus Type 2; Crestor, Rosuvastatin; LDL Cholesterol; Observational
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine in DM II patients the efficacy of Crestor in obtaining the new European LDL cholesterol guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus Type 2, LDL-C > 2,5 mmol/l, no cholesterol lowering medication used last 3 months, starts with Crestor 10 mg, permission to use patient data by AZ

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes Mellitus Type 2
Sampling Method: Probability Sample
Enrollment: 2500
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Astra Zeneca, Study Director — AstraZeneca
Locations (222):
- Netherlands (222):
  - Research Site, 's Gravenmoer
  - Research Site, 's-Hertogenbosch
  - Research Site, Aalten
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Alphen aan den Rijn
  - Research Site, Amersfoort
  - Research Site, Ammerzoden
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Amsterdam-Zuidoost
  - Research Site, Andijk
  - Research Site, Apeldoorn
  - Research Site, Arcen
  - Research Site, Arkel
  - Research Site, Arnhem
  - Research Site, Assen
  - Research Site, Baard
  - Research Site, Baarle-Nassau
  - Research Site, Baflo
  - Research Site, Beek en Donk
  - Research Site, Benningbroek
  - Research Site, Bergeijk
  - Research Site, Bergen op Zoom
  - Research Site, Best
  - Research Site, Beverwijk
  - Research Site, Bilthoven
  - Research Site, Blaricum
  - Research Site, Bocholtz
  - Research Site, Boekel
  - Research Site, Boxtel
  - Research Site, Breda
  - Research Site, Brunssum
  - Research Site, Budel
  - Research Site, Burgum
  - Research Site, Bussum
  - Research Site, Callantsoog
  - Research Site, Capelle aan den IJssel
  - Research Site, Castricum
  - Research Site, Coevorden
  - Research Site, Cuijk
  - Research Site, Damwoude
  - Research Site, Delft
  - Research Site, Delfzijl
  - Research Site, Den Helder
  - Research Site, Deurne
  - Research Site, Dieren
  - Research Site, Dirksland
  - Research Site, Doesburg
  - Research Site, Doetinchem
  - Research Site, Dokkum
  - Research Site, Doorn
  - Research Site, Drachten
  - Research Site, Duiven
  - Research Site, Echt
  - Research Site, Ede Gld
  - Research Site, Eemnes
  - Research Site, Eersel
  - Research Site, Egmond aan den Hoef
  - Research Site, Eibergen
  - Research Site, Eindhoven
  - Research Site, Elim
  - Research Site, Emmeloord
  - Research Site, Emmen
  - Research Site, Enkhuizen
  - Research Site, Enschede
  - Research Site, Exloo
  - Research Site, Garderen
  - Research Site, Geldrop
  - Research Site, Geleen
  - Research Site, Goes
  - Research Site, Goirle
  - Research Site, Gorinchem
  - Research Site, Groningen
  - Research Site, Grootebroek
  - Research Site, Haarlem
  - Research Site, Hapert
  - Research Site, Hardenberg
  - Research Site, Haren
  - Research Site, Harskamp
  - Research Site, Havelte
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Heeswijk-Dinther
  - Research Site, Heiloo
  - Research Site, Hellevoetsluis
  - Research Site, Helmond
  - Research Site, Hengelo Ov
  - Research Site, Hillegom
  - Research Site, Hoogeveen
  - Research Site, Hoogvliet
  - Research Site, Hoorn
  - Research Site, Horst
  - Research Site, Houten
  - Research Site, Huizen
  - Research Site, Hulst
  - Research Site, IJmuiden
  - Research Site, Joure
  - Research Site, Kilder
  - Research Site, Klazienaveen
  - Research Site, Koekange
  - Research Site, Lage Mierde
  - Research Site, Landgraaf
  - Research Site, Landsmeer
  - Research Site, Laren Nh
  - Research Site, Leek
  - Research Site, Leersum
  - Research Site, Leeuwarden
  - Research Site, Leiden
  - Research Site, Lemmer
  - Research Site, Leusden
  - Research Site, Lichtenvoorde
  - Research Site, Lieshout
  - Research Site, Limmen
  - Research Site, Lisse
  - Research Site, Lunteren
  - Research Site, Maarn
  - Research Site, Maarssen
  - Research Site, Maastricht
  - Research Site, Meerlo
  - Research Site, Melick
  - Research Site, Meppel
  - Research Site, Milsbeek
  - Research Site, Montfoort
  - Research Site, Moordrecht
  - Research Site, Musselkanaal
  - Research Site, Naarden
  - Research Site, Neede
  - Research Site, Nibbixwoud
  - Research Site, Nieuw-Buinen
  - Research Site, Nieuwdorp Zld
  - Research Site, Nieuwe Pekela
  - Research Site, Nieuwegein
  - Research Site, Nieuwendijk Nb
  - Research Site, Nijverdal
  - Research Site, Noord-Scharwoude
  - Research Site, Noordscheschut
  - Research Site, Noordwijk Zh
  - Research Site, Nunspeet
  - Research Site, Oegstgeest
  - Research Site, Oldenzaal
  - Research Site, Oost West en Middelbeers
  - Research Site, Oosterhout Nb
  - Research Site, Oss
  - Research Site, Oud-Beijerland
  - Research Site, Oude Pekela
  - Research Site, Oudega Gem Smallingerlnd
  - Research Site, Oudorp Nh
  - Research Site, Pijnacker
  - Research Site, Poeldijk
  - Research Site, Poortvliet
  - Research Site, Purmerend
  - Research Site, Ridderkerk
  - Research Site, Rijnsburg
  - Research Site, Rijsbergen
  - Research Site, Rijssen
  - Research Site, Rockanje
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Rozenburg Zh
  - Research Site, Schoonhoven
  - Research Site, Sint Willebrord
  - Research Site, Sint-Oedenrode
  - Research Site, Sliedrecht
  - Research Site, Sneek
  - Research Site, Sommelsdijk
  - Research Site, Son
  - Research Site, Spijkenisse
  - Research Site, Stadskanaal
  - Research Site, Steenbergen Nb
  - Research Site, T Zand Nh
  - Research Site, Ten Boer
  - Research Site, Ter Aar
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Tuitjenhorn
  - Research Site, Uden
  - Research Site, Ulft
  - Research Site, Usquert
  - Research Site, Utrecht
  - Research Site, Valkenswaard
  - Research Site, Veenendaal
  - Research Site, Veghel
  - Research Site, Velden
  - Research Site, Veldhoven
  - Research Site, Venlo
  - Research Site, Venray
  - Research Site, Vlaardingen
  - Research Site, Vledder
  - Research Site, Vlijmen
  - Research Site, Voerendaal
  - Research Site, Volendam
  - Research Site, Voorburg
  - Research Site, Voorhout
  - Research Site, Voorschoten
  - Research Site, Vries
  - Research Site, Vught
  - Research Site, Waalre
  - Research Site, Wamel
  - Research Site, Warmond
  - Research Site, Warnsveld
  - Research Site, Weert
  - Research Site, Westerhaar-vriezenv Wijk
  - Research Site, Westervoort
  - Research Site, Wijchen
  - Research Site, Wildervank
  - Research Site, Winschoten
  - Research Site, Winterswijk
  - Research Site, Wognum
  - Research Site, Zeewolde
  - Research Site, Zeist
  - Research Site, Zevenhuizen Gn
  - Research Site, Zoetermeer
  - Research Site, Zuidhorn
  - Research Site, Zuidlaren
  - Research Site, Zutphen
  - Research Site, Zwaag
  - Research Site, Zwaagwesteinde
  - Research Site, Zwijndrecht
  - Research Site, Zwolle